CLINICAL TRIAL: NCT04956445
Title: Collection of SARS CoV-2 (COVID-19) Virus Secretions and Serum for Countermeasure Development
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tulane University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-396
Record Dates: First submitted 2021-06-18; First posted 2021-07-09 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Data registry; Convalescent plasma; Post COVID-19; Post acute sequelae of COVID-19
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigators are collecting blood, plasma, urine, stool, nasal swab, saliva and tears collection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population 1: Once a positive diagnosis of COVID-19 has been made in the clinical setting, the clinical team caring for the patient will ask the patient / family whether they would be willing to be contacted by the study team about the study. If so, a trained member of the study team will describe the study in person or by telephone. Community members who see the study flyer will also be able to reach out to the study team to learn more about the study and to find out if they meet eligibility criteria. If the eligible patient / legally authorized representative / legal guardian would like to participate. The verbal informed consent / verbal HIPAA, assent, and/or parental permission (as appropriate) will then be obtained in person.
- Population 2: Persons with a history of past (>14 days ago) diagnosis of COVID-19 infection will be invited to participate in this study. In addition, persons who have had significant exposure to a patient with COVID-19 (contact at a distance of less than 6 feet without personal protective equipment) and have remained asymptomatic for 14 days following exposure will be recruited. Candidates will be identified through initial enrollment in Population 1, or by clinicians who have been informed of the study but are not part of the study team. Then, the clinical care team will ask the patient if he/she is willing to be contacted by the study team. Community members who see the study flyer or are otherwise informed of the study will also be able to reach out to the study team. Additionally, individuals with no defined past COVID-19 infection, but the potential to have been exposed to, and mounted antibodies against, COVID-19 will also be enrolled in Population 2 for this study.

SUMMARY:
Collection of SARS-COV-2 Secretions and Serum for Countermeasure Development (aka ClinSeqSer) is an observational study to understand natural history of SARS-COV-2 infections among special populations and characterise post-covid morbidity through immune response, virus genome sequencing, cytokine response, and virus shedding. Given the descriptions of infection course of patients over the outbreak of 2003 (SARS-Cov01) and since January 2019 in China and Europe, and now worldwide:

1. Acutely infected patients shed virus that could be of major interest to characterize (viral quantification, characterization of virus shedding -of infective and of non-infective virus) the former reflecting/predictive of severity of disease and the latter reflecting extent/source of contagiosity.
2. Convalescent infected patients develop a specific anti-virus antibody response that is (likely) protective and therefore suits the preliminary requirement for the potential benefits of the convalescent patient plasma therapeutic infusion approach. In addition, long term effects of COVID-19 commonly known as long-haulers remains clinically unclear.

Thousands of patients have now been diagnosed with COVID-19 in Louisiana (444,000 cases, 10,122 deaths, 2.2% mortality in Louisiana (LA), as of March 2021), and numerous patients are now also complaining of post-acute sequelae of SARS-CoV-2 (PASC). The investigators want to further clarify questions surrounding rational confinement duration and therapeutic approach by collecting plasma of convalescent patients to identify optimal antibody titer by ELISA, specificity of naturally occurring inflammatory (protein/antibody and RNA) response, and possibly test in vitro antibody neutralization activity.

DETAILED DESCRIPTION:
The investigators are proposing two strategies to help mitigate COVID-19:

1. Establish active data registry for infected patients, which includes both sequence of viral isolate and clinical course. The purpose of this would be to determine whether sequences are evolving, which might affect planned countermeasures, and to evaluate which comorbidities/concurrent medications/clinical findings are the highest predictors for risk. This could allow us to better target screening and triage efforts, and potentially discontinue/substitute out medications that are worsening infection. For example, if diabetics confirm to be a particularly high risk they should potentially receive more rigorous screening, earlier admission, earlier medication optimization. For another example, there is some concern that patients with hypertension on angiotensin receptor blocking agents may have enhanced expression of Angiotensin Converting Enzyme (ACE-2), the entry receptor for SARS-CoV-2. If the investigators can confirm whether patients on Angiotensin Receptor Blocker (ARBs) have severe outcomes, this would justify the potential switch to alternate agents. Collect serum/plasma from convalescent patients. Patients who have been diagnosed with COVID-19 and have recovered (>14 days since diagnosis) or individuals with no defined past COVID-19 infection, but the potential to have been exposed to (and mounted antibodies against) COVID-19 will provide a sample of whole blood, as well as other samples.
2. Determine long-term sequelae and pulmonary-related health outcomes for infected patients with COVID-19. Patients who survive infection with SARS Cov-2 are at risk of physical and psychological complications of lung injury. The investigators aim to determine the long-term sequelae of this infection. This would allow the investigators to better understand the long-term health impacts (physiological, functional, and quality-of-life) of this disease. Specifically, they aim to 1) conduct a systematic study of subjects post-COVID in order to determine which part(s) of that morbidity (clinical and laboratory) is caused by COVID, and 2) Identify predictors of post-COVID morbidity, including any protective role of treatments used during acute infection, and identify biomarkers (virus and host) that might be associated with severity/duration of the post-COVID syndrome. Overall, the investigators aim to define the entity of post-COVID morbidity, or post-acute sequelae of SARS-CoV-2 (PASC) so that they can then begin to explore methods to treat, and, ideally, prevent this morbidity.

The investigators are expanding the criteria for inclusion in this study to other viruses in order to

1. Develop a comparator group to determine whether immunomodulation induced by SARS CoV-2 differs from other respiratory viruses,
2. Prepare for both routine seasonal and potential future influenza pandemic, which has been an ongoing concern for years now, and
3. Expand their ability to monitor for potential intermixing of seasonal coronaviruses and SARS CoV-2, which could impact diagnostic tests for both.

ELIGIBILITY:
Population 1:

Inclusion Criteria:

1. Positive diagnostic test for COVID-19, influenza A or B virus, non COVID-19 coronavirus, parainfluenza virus, rhinovirus, adenovirus, or metapneumovirus
2. Patient or legally authorized representative has provided verbal consent / verbal HIPAA (or parental permission form and assent form, as appropriate)

Exclusion Criteria:

* None

Population 2:

Inclusion Criteria:

1. Positive diagnostic test for COVID-19 >14 days prior, OR potential to have been exposed to (and mounted antibodies against) COVID-19, OR positive diagnostic test for influenza A or B virus, non COVID-19 coronavirus, parainfluenza virus, rhinovirus, adenovirus, or metapneumovirus
2. Patient or legally authorized representative has signed informed consent (or parental permission form and assent form, as appropriate)

Exclusion Criteria:

Patients with the following criteria:

* Aged under 6 months old
* Anemia (Hgb <7)
* Platelet <80

Ages: 6 Months to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population 1: Infected patients
  Once a positive diagnosis of COVID-19 has been made in the clinical setting, the clinical team caring for the patient will ask the patient / family whether they would be willing to be contacted by the study team about the study.
  Population 2: Convalescent patients
  Persons with a history of past (>14 days ago) diagnosis of COVID-19 infection will be invited to participate in this study. In addition, persons who have had a significant exposure to a patient with COVID-19 (contact at distance of less than 6 feet without personal protective equipment) and have remained asymptomatic for 14 days following exposure will be recruited.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
COVID-19 clinically severe vs non severe cases | 2 Years
  To determine the clinical and laboratory risk factors which lead to severe vs non-severe COVID-19 clinical course in ambulatory patients.
  Severe COVID-19 cases defined as death or hospitalized on invasive mechanical ventilation or Extracorporeal membrane oxygenation (ECMO).
  Non-severe COVID-19 cases defined as hospitalized on non-invasive ventilation or high flow oxygen devices or requiring low flow supplemental oxygen (less than 15L) or not requiring supplemental oxygen, requiring ongoing medical care or no longer requires on going medical care or not hospitalized.
Post-COVID symptoms onset at 3 months | 3 Months
  The proportion (in percentage) of the study cohort exhibiting post-COVID symptoms after recovering from COVID-19 at 3 months from initial date of symptom onset. Post-COVID symptoms which are all new since COVID infection are fatigue, tiredness or exhaustion, muscle aches/muscle pains, pain in joints, problems in sleep, forgetfulness/memory problems, difficulty thinking or concentrating, dizziness or fainting, fever, headache, nausea or abdominal pain, diarrhea, runny nose, sore throat, cough, shortness of breath/abnormal breathing, loss of smell, loss of taste, and inability to walk.

SECONDARY OUTCOMES:
Post-COVID symptoms onset at 6 months | 6 months
  The proportion (in percentage) of the study cohort exhibiting post-COVID symptoms after recovering from COVID-19 at 6 months from initial date of symptom onset. Post-COVID symptoms which are all new since COVID infection are fatigue, tiredness or exhaustion, muscle aches/muscle pains, pain in joints, problems in sleep, forgetfulness/memory problems, difficulty thinking or concentrating, dizziness or fainting, fever, headache, nausea or abdominal pain, diarrhea, runny nose, sore throat, cough, shortness of breath/abnormal breathing, loss of smell, loss of taste, and inability to walk.
Post-COVID symptoms onset at 9 months | 9 months
  The proportion (in percentage) of the study cohort exhibiting post-COVID symptoms after recovering from COVID-19 at 9 months from initial date of symptom onset. Post-COVID symptoms which are all new since COVID infection are fatigue, tiredness or exhaustion, muscle aches/muscle pains, pain in joints, problems in sleep, forgetfulness/memory problems, difficulty thinking or concentrating, dizziness or fainting, fever, headache, nausea or abdominal pain, diarrhea, runny nose, sore throat, cough, shortness of breath/abnormal breathing, loss of smell, loss of taste, and inability to walk.
Post-COVID symptoms onset at 12 months | 12 months
  The proportion (in percentage) of the study cohort exhibiting post-COVID symptoms after recovering from COVID-19 at 12 months from initial date of symptom onset. Post-COVID symptoms which are all new since COVID infection are fatigue, tiredness or exhaustion, muscle aches/muscle pains, pain in joints, problems in sleep, forgetfulness/memory problems, difficulty thinking or concentrating, dizziness or fainting, fever, headache, nausea or abdominal pain, diarrhea, runny nose, sore throat, cough, shortness of breath/abnormal breathing, loss of smell, loss of taste, and inability to walk.
Post-COVID symptoms onset at 15 months | 15 months
  The proportion (in percentage) of the study cohort exhibiting post-COVID symptoms after recovering from COVID-19 at 15 months from initial date of symptom onset. Post-COVID symptoms which are all new since COVID infection are fatigue, tiredness or exhaustion, muscle aches/muscle pains, pain in joints, problems in sleep, forgetfulness/memory problems, difficulty thinking or concentrating, dizziness or fainting, fever, headache, nausea or abdominal pain, diarrhea, runny nose, sore throat, cough, shortness of breath/abnormal breathing, loss of smell, loss of taste, and inability to walk.
Post-COVID symptoms onset at 18 months | 18 months
  The proportion (in percentage) of the study cohort exhibiting post-COVID symptoms after recovering from COVID-19 at 18 months from initial date of symptom onset. Post-COVID symptoms which are all new since COVID infection are fatigue, tiredness or exhaustion, muscle aches/muscle pains, pain in joints, problems in sleep, forgetfulness/memory problems, difficulty thinking or concentrating, dizziness or fainting, fever, headache, nausea or abdominal pain, diarrhea, runny nose, sore throat, cough, shortness of breath/abnormal breathing, loss of smell, loss of taste, and inability to walk.
Post-COVID symptoms onset at 21 months | 21 months
  The proportion (in percentage) of the study cohort exhibiting post-COVID symptoms after recovering from COVID-19 at 21 months from initial date of symptom onset. Post-COVID symptoms which are all new since COVID infection are fatigue, tiredness or exhaustion, muscle aches/muscle pains, pain in joints, problems in sleep, forgetfulness/memory problems, difficulty thinking or concentrating, dizziness or fainting, fever, headache, nausea or abdominal pain, diarrhea, runny nose, sore throat, cough, shortness of breath/abnormal breathing, loss of smell, loss of taste, and inability to walk.
Post-COVID symptoms onset at 24 months | 24 months
  The proportion (in percentage) of the study cohort exhibiting post-COVID symptoms after recovering from COVID-19 at 24 months from initial date of symptom onset. Post-COVID symptoms which are all new since COVID infection are fatigue, tiredness or exhaustion, muscle aches/muscle pains, pain in joints, problems in sleep, forgetfulness/memory problems, difficulty thinking or concentrating, dizziness or fainting, fever, headache, nausea or abdominal pain, diarrhea, runny nose, sore throat, cough, shortness of breath/abnormal breathing, loss of smell, loss of taste, and inability to walk.

CONTACTS AND LOCATIONS:
Overall Officials: Dahlene Fusco, MD, PhD, Principal Investigator — Tulane University School of Medicine
Locations (2):
- United States (2):
  - Tulane University Medical Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana